CLINICAL TRIAL: NCT02212509
Title: Functional Recovery After Cardiac Surgery : Does Delirium and Calorie Intake Matter?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201203074RIC
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Disorder; Heart, Functional, Postoperative, Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aims of the cohort study is to describe the rates of 30-day surgical complication, functional decline, frailty and one-year mortality for patients experienced cardiac surgery and to delineate the trajectory of functional capacity 1 year after surgery for the patients. It also will test whether the trajectory of functional varied significantly according to delirium status and its type over the follow-up period and examine the patients' postsurgical actual caloric/protein/fluid intake in relation to the functional capacity within 3 months after surgery as well as evaluate whether activity levels, dietary diversity, and depressive symptoms at 3,6, and 12 months affect patient outcome.

DETAILED DESCRIPTION:
In Taiwan, 54.2% of cardiac surgical procedures in 2010 were performed on older patients (≧65 years) with higher rates of surgical complications, functional decline, and even death reported. Despite the large number of older patients undergoing cardiac surgery with the goal of improving functional capacity, the literature in this area is limited. Specifically, there is little information about the functional outcomes 1 year after cardiac surgery for older patients.

A prospective, longitudinal cohort study will be conducted to assess and follow patients aged 65 years and older who undergoing elective or non-elective cardiac surgery for one year after surgery. All patients on the cardio-surgical wards of 5A, 5B, and 5CVI at National Taiwan University Hospital will be screened for eligibility. Every patient ≧65 years admitted for cardiac surgery will be approached and invited to participate. This cohort study aims to 1)describe the rates of 30-day surgical complication, functional decline, frailty, and one-year mortality for older patients underwent cardiac surgery; 2) delineate the rajectory of functional capacity 1 year after surgery for these patients; 3) test whether the trajectory of functional capacity varied significantly according to delirium status and its type over the one-year follow-up period; 4)examine patients' postsurgical actual caloric/protein/fluid intake in relation to the functional capacity within 3 months after surgery; and 5) evaluate hether activity levels, dietary diversity, and depressive symptoms at 3, 6, and 12 months affect patient outcomes. Estimated 236 participants will be enrolled to ensure the power of study.

Data will be analyzed using the SAS package. The Generalized Estimating Equation (GEE) will be performed to identify the risk factors and to delineate the trajectory of functional capacity 1 year after cardiac surgery for older patients. The findings will add to the development of nursing intervention program to promote functional recovery for older patients after cardiac surgery

ELIGIBILITY:
Inclusion Criteria:

* patients over 20 years old
* admitted for elective or non-elective cardiac surgery

Exclusion Criteria:

* incapable of verbal communication
* sensory impairment
* intubation or respiratory isolation
* patients with critical condition or coma

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients on the cardio-surgical wards
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
physical activity function | admission and 1 year after surgery

SECONDARY OUTCOMES:
mortality | 1 year after surgery

OTHER OUTCOMES:
30 days surgical complication | 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan